CLINICAL TRIAL: NCT07023471
Title: Effect of an Artificial Intelligence-assisted Colonoscopy on Adenoma Miss Rate of Trainee-performed Colonoscopy: A Four-group Randomized Controlled Tandem Colonoscopy Study
Brief Title: Artificial Intelligence-assisted Colonoscopy, Tandem Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nonthalee Pausawasdi, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Si299/2025
Record Dates: First submitted 2025-06-07; First posted 2025-06-17 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Artificial Intelligence (AI); Colonoscopy Education; Adenoma Colon Polyp
Keywords: Adenoma miss rate; Artificial intelligence; colonoscopy; tandem colonoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Trainee --> expert) (Placebo Comparator): The expert endoscopist insert to cecum in both passes. First pass: Trainee withdraw colonoscopy without AI. The polyps detected can be removed as suitable. The pathology for polyp will be sent.
  Second pass: Expert withdraw colonoscopy without AI. The polyps detected (which is missed from the first pass) can be removed as suitable. The pathology for polyp will be sent.
  Interventions: Device: Group A (Trainee --> expert)
- Group B (Trainee +AI --> expert) (Other): The expert endoscopist insert to cecum in both passes. First pass: Trainee withdraw colonoscopy with AI. The polyps detected can be removed as suitable. The pathology for polyp will be sent.
  Second pass: Expert withdraw colonoscopy without AI. The polyps detected (which is missed from the first pass) can be removed as suitable. The pathology for polyp will be sent.
  Interventions: Device: Group B (Trainee +AI --> expert)
- Group C (Trainee --> expert + AI) (Other): The expert endoscopist insert to cecum in both passes. First pass: Trainee withdraw colonoscopy without AI. The polyps detected can be removed as suitable. The pathology for polyp will be sent.
  Second pass: Expert withdraw colonoscopy with AI. The polyps detected (which is missed from the first pass) can be removed as suitable. The pathology for polyp will be sent.
  Interventions: Device: Group C (Trainee --> expert + AI)
- Group D (Trainee + AI --> expert + AI) (Other): The expert endoscopist insert to cecum in both passes. First pass: Trainee withdraw colonoscopy with AI. The polyps detected can be removed as suitable. The pathology for polyp will be sent.
  Second pass: Expert withdraw colonoscopy with AI. The polyps detected (which is missed from the first pass) can be removed as suitable. The pathology for polyp will be sent.
  Interventions: Device: Group D (Trainee + AI --> expert + AI)

INTERVENTIONS:
Device: Group A (Trainee --> expert) — The expert endoscopist insert to cecum in both passes. First pass: Trainee withdraw colonoscopy (white-light mode) without AI. The polyps detected can be removed as suitable. The pathology for polyp will be sent. Second pass: Expert withdraw colonoscopy (white-light mode) without AI. The polyps detected (which is missed from the first pass) can be removed as suitable. The pathology for polyp will be sent.
  Arms: Group A (Trainee --> expert)
Device: Group B (Trainee +AI --> expert) — The expert endoscopist insert to cecum in both passes. First pass: Trainee withdraw colonoscopy with AI. The polyps detected can be removed as suitable. The pathology for polyp will be sent. Second pass: Expert withdraw colonoscopy (white-light mode) without AI. The polyps detected (which is missed from the first pass) can be removed as suitable. The pathology for polyp will be sent.
  Artificial intelligent (AI) assisted colonoscopy; ENdoscopy as AI-powered Device (ENAD) ENAD system (ENdoscopy as AI-powered Device, AINEX Corporation, Seoul, South Korea) is the system using CADe system (Computer-aided detection) which developed from 66,397 images and 8,756 polyps via deep learning-based object detection algorithm (YOLOv4) . It was validated by 15,753 images of polyp from 80 colonoscopy videos and 90,144 images of non-polyps from 50 colonoscopy videos. This system decreases false positive rate from 3.2% to 0.6% and increases sensitivity from 86.4% to 87.1%.
  Arms: Group B (Trainee +AI --> expert)
Device: Group C (Trainee --> expert + AI) — The expert endoscopist insert to cecum in both passes. First pass: Trainee withdraw colonoscopy (white-light mode) without AI. The polyps detected can be removed as suitable. The pathology for polyp will be sent. Second pass: Expert withdraw colonoscopy with AI. The polyps detected (which is missed from the first pass) can be removed as suitable. The pathology for polyp will be sent.
  Artificial intelligent (AI) assisted colonoscopy; ENdoscopy as AI-powered Device (ENAD) ENAD system (ENdoscopy as AI-powered Device, AINEX Corporation, Seoul, South Korea) is the system using CADe system (Computer-aided detection) which developed from 66,397 images and 8,756 polyps via deep learning-based object detection algorithm (YOLOv4) . It was validated by 15,753 images of polyp from 80 colonoscopy videos and 90,144 images of non-polyps from 50 colonoscopy videos. This system decreases false positive rate from 3.2% to 0.6% and increases sensitivity from 86.4% to 87.1%.
  Arms: Group C (Trainee --> expert + AI)
Device: Group D (Trainee + AI --> expert + AI) — The expert endoscopist insert to cecum in both passes. First pass: Trainee withdraw colonoscopy with AI. The polyps detected can be removed as suitable. The pathology for polyp will be sent. Second pass: Expert withdraw colonoscopy with AI. The polyps detected (which is missed from the first pass) can be removed as suitable. The pathology for polyp will be sent.
  Artificial intelligent (AI) assisted colonoscopy; ENdoscopy as AI-powered Device (ENAD) ENAD system (ENdoscopy as AI-powered Device, AINEX Corporation, Seoul, South Korea) is the system using CADe system (Computer-aided detection) which developed from 66,397 images and 8,756 polyps via deep learning-based object detection algorithm (YOLOv4) . It was validated by 15,753 images of polyp from 80 colonoscopy videos and 90,144 images of non-polyps from 50 colonoscopy videos. This system decreases false positive rate from 3.2% to 0.6% and increases sensitivity from 86.4% to 87.1%.
  Arms: Group D (Trainee + AI --> expert + AI)

SUMMARY:
The goal of this clinical trial is to evaluate effect of artifial intelligent (AI) system, Endoscopy as AI-powered Device (ENAD) on adenoma miss rate from colonoscopy underwent by trainee endoscopist. It will also evaluate effect of AI on adenoma and polyp detection rate from colonoscopy underwent by trainee endoscopist. The main questions it aims to answer are:

• Does AI-system lower adenoma miss rate in colonoscopy underwent by trainee endoscopist?

Researchers will do the tandem colonoscopy and devided the participant in 4 groups as follows:

A. First pass: trainee; Second pass: expert B. First pass: trainee + AI; Second pass: expert C. First pass: trainee; Second pass: expert + AI D. First pass: trainee+AI; Second pass: expert+AI Participants will take bowel preparation in split dose regimen and nothing per oral for 4 hours. They will underwent colonoscopy as above, with sedation by anesthesiologist. Details on qualities of colonoscopy, polyps detection and pathology results will be recorded.

DETAILED DESCRIPTION:
Colon cancer accounts for one of the most common cancer worldwide and also cancer-related death. Colonoscopy is accepted to be an effective tool in colon cancer screening since the polypectomy of small adenoma can prevent colon cancer. Missed adenoma is one of the causes of interval cancer between routine colonoscopy screening. Nonvisualization is the cause of missed adenoma during colonoscopy. Artificial intelligence (AI)-assisted colonoscopy was superior then routine colonoscopy from parallel study and tandem study. Previous studies often used one same endoscopist in doing tandem colonoscopy which may still have bias. Only one previous study designed to use trainee endoscopist in the first pass and expert endoscopist in the second pass, some subgroups used AI-assisted. The result revealed the lower of adenoma miss rate (AMR) in AI-assisted colonoscopy in the first pass. This study designed to evaluate AMR of AI-assisted colonoscopy in trainee endoscopist compared to expert endoscopist, the trainee will do colonoscopy in the first pass (with or without AI) and the expert will do colonoscopy in the second pass (with or without AI). The present study aimed to evaluate effect of AI-assisted colonoscopy in trainee endoscopist.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 - 85 years old
* Appointment for colonoscopy for colorectal cancer screening

Exclusion Criteria:

* Previous history of bowel obstruction or perforation
* Presence of coagulopathy (Prothrombin time >, = 3 second ULN; Platelet < 50,000)
* Previously diagnosed with inflammatory bowel disease or polyposis syndrome
* Pregnancy or lactation
* Severe comorbities or American Society of Anesthesiologist classification >, = 3
* Unable to sign informed consent

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adenoma miss rate | Untill the end of procedure
  Compare adenoma miss rate (AMR) in each groups including Non-AI/ Non-AI, Non-AI/ AI, AI/ Non-AI, and AI/ AI

SECONDARY OUTCOMES:
Polyp miss rate | Untill the end of the procedure
  Compare polyp miss rate (PMR) in each groups
Adenoma detection rate of colonoscopy underwent by the trainee | Untill the end of procedure of first pass which will be done by trainee
  Compare adenoma detection rate (ADR) of colonoscopy underwent by trainee with or without AI

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The investigators are willing to provide our data to researchers who require it. For example, those who want to do systematic review and meta-analysis.
Supporting Information: Study Protocol
Time Frame: Other researchers can contact us anytime
Access Criteria: The investigators will provide our protocol and/or data upon request.